CLINICAL TRIAL: NCT04780334
Title: Rapid Detection of COVID-19 by Portable and Connected Biosensor : Biological Proof of Concept
Acronym: COR-DIAL-S
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0063; 2021-A00387-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-03-02; First posted 2021-03-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV Infection; Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — nasopharyngeal swab and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive diagnosis of SARS-CoV-2: 100 patients with a positive diagnosis of SARS-CoV-2
  Interventions: Diagnostic Test: COVID-19 RT-PCR; Diagnostic Test: Biosensor
- Negative diagnosis of SARS-CoV-2: 100 patients with a negative diagnosis of SARS-CoV-2 defined by the gold standard by the medical team
  Interventions: Diagnostic Test: COVID-19 RT-PCR; Diagnostic Test: Biosensor

INTERVENTIONS:
Diagnostic Test: COVID-19 RT-PCR — Nasopharyngeal swabs for COVID-19 RT-PCR
Diagnostic Test: Biosensor — Portable and Connected Biosensor viral

SUMMARY:
The main objective of this CorDial-S proof-of-concept study is to evaluate the ability to detect COVID-19 infection in nasopharyngeal swabs with CorDial-S and compare it to the PCR technique currently in use. Saliva analysis will be the subject of secondary analysis.

The CorDial-S medical device could allow the specimens to be analyzed using a small portable device and the results to be returned in minutes to the medical team and the patient, and communicated in real time with a telemedicine and remote monitoring system to the health authorities to allow the necessary protective, containment and therapeutic management measures to be put in place if necessary.

The benefits would be

1. greater sensitivity
2. a great speed because 8tests could be performed at the same time with a result in a few minutes
3. a very high specificity at least equivalent to PCR.

This new diagnostic strategy could become extremely valuable in the fight against COVID-19, especially in the case of very long-term persistence and incomplete vaccination of the French and foreign population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female or child without age limit
* Admitted to a Reference Health Establishment (RHS) in an emergency unit, hospitalization or intensive care unit for suspicion of SARS-CoV-2 infection regardless of clinical presentation and degree of severity.
* Patient to be diagnosed by PCR test on nasopharyngeal swab.
* Social insured

Exclusion Criteria:

* Refusal of the person to participate (collection of information, second use of his sample, collection of saliva by spitting)
* Pregnant and breastfeeding women
* Protected Majors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to a Reference Health Establishment for suspicion of SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of CorDial-S based on the first nasopharyngeal swab taken on patient admission, compared to the final positive or negative diagnosis of COVID-19 by the medical team | at patient admission (Baseline)

SECONDARY OUTCOMES:
Cohen's Kappa Coefficient for concordance for the diagnosis of CoV-2-SARS between PCR and CorDial-S based on nasopharyngeal swabs taken at patient admission. | at patient admission (Baseline)
Sensitivity and specificity of CorDial-S based on the first saliva sample taken at patient admission compared to the final positive or negative diagnosis of COVID-19 by the medical team. | at patient admission (Baseline)
Cohen's Kappa Coefficient for concordance for the diagnosis of CoV-2-SARS between PCR and CorDial-S based on saliva samples taken at patient admission. | at patient admission (Baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Enagnon Kazali ALIDJINOU, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France